CLINICAL TRIAL: NCT03686176
Title: Virtual Reality During Procedures in Pediatric Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Coronavirus (COVID-19)-related pause on all clinical research studies.
Sponsor: Johns Hopkins University (Other)
Collaborators: The Thomas Wilson Sanitarium for Children of Baltimore City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00161331
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Results first posted 2020-07-28 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Virtual Reality; Pediatrics

STUDY DESIGN:
Intervention Model Description: randomized, unblinded, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (Study Group) (Experimental): In this arm, patients will receive support from child life specialists plus may use virtual reality simulation goggles during a qualifying medical procedure.
  Interventions: Other: Virtual Reality
- Active Control Group (No Intervention): In this arm, patients will receive standard of care with child life specialists plus distraction of the child's choosing, during a qualifying medical procedure.
- External Control (Reference Group) (No Intervention): No virtual reality and no child life specialists; no standardized or formal form of support.

INTERVENTIONS:
Other: Virtual Reality — A child life specialist will fit the patient with the goggles, select a game, and initiate play once the medical procedure begins.
  Other Names: Oculus Go
  Arms: Virtual Reality Group (Study Group)

SUMMARY:
This stratified, randomized, controlled trial compared coping and distress between child life supported virtual reality engagement and child life support during painful procedures in the pediatric emergency department.

DETAILED DESCRIPTION:
Pediatric emergency rooms and hospitals are anxiety provoking and often painful places for pediatric patients and families. Children of all ages present to the Johns Hopkins emergency room and are admitted to the hospital for a wide range of medical conditions, many of which require medical interventions. Many of these interventions are the source of anxiety and pain, including burn debridement or dressing changes, laceration repair, or intravenous (IV) line placement. The standard of care to reduce pain and improve coping during pediatric procedures ranges from no intervention to support from child life specialists.

As an adjunct to the existing methods of promoting comfort during painful procedures, non-invasive virtual reality (VR) therapy is showing promise as a means of distraction and coping with various medical procedures. The user is transported into a relaxing/distracting VR environment that diverts user's attention away from pain and anxiety. VR has demonstrated efficacy in the reduction of pain and anxiety experienced by individuals undergoing anxiety and pain inducing procedures.While there is early data from small or narrow populations that show some improvement in pain and anxiety with VR use during pediatric procedures, some studies show no improvement. No studies to date have used objective outcome measures of coping, which may be more clinically meaningful.

The investigators propose to fill this gap in the literature with a randomized, controlled, un-blinded study of coping and distress between virtual reality engagement and child life support in pediatric patients undergoing painful medical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients requiring painful or anxiety inducing procedures:

   * Burn debridement
   * Burn dressing change
   * Lactation repair
   * Intravenous (IV) line placement or phlebotomy (blood draw)
   * Abscess incision and drainage
   * Fracture reduction and/or cast placement
   * Implanted central venous port placement accessing
   * Skin biopsies
2. Subjects ages 7 to 26 years of age (age 26 is the upper limit treated at JHCC) Ages were chosen based on that previously published in the literature on pediatric patients with VR.

Exclusion Criteria:

* Patients with a known history of a seizure disorder.
* Patients with an active infection, burn, or trauma that interferes with the mask placement, and may include involvement of the periorbital skin, eyes, nasal bridge, external ear, and/or scalp or hair.
* Patients with Blindness.
* Developmental delay significant enough to interfere with the subject's ability to participate in the session, including autism spectrum disorders.
* Patients with active psychosis or exhibit signs of active intoxication.
* Known history of severe motion sickness
* Medical urgency (at the medical providers' discretion)
* Non-verbal children
* Children or parents/legal guardians who are non-English speakers

Ages: 7 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Therese Canares, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Children's Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Canares T, Parrish C, Santos C, Badawi A, Stewart A, Kleinman K, Psoter K, McGuire J. Pediatric Coping During Venipuncture With Virtual Reality: Pilot Randomized Controlled Trial. JMIR Pediatr Parent. 2021 Jul 28;4(3):e26040. doi: 10.2196/26040. PMID 34319249
- [Derived] Canares TL, Parrish C, Santos C, Badawi A, Stewart A, Kleinman K, Psoter KJ, McGuire JF. Resource Use During Pediatric Venipuncture With Virtual Reality: Secondary Analysis of a Randomized Controlled Pilot Trial. Hosp Pediatr. 2021 Jul;11(7):775-778. doi: 10.1542/hpeds.2020-003822. Epub 2021 Jun 14. PMID 34127486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the pediatric emergency department (PED) at an urban, tertiary care children's hospital.
Groups:
- Virtual Reality Group (Study Group): In this arm, patients will receive standard of care plus may use virtual reality simulation goggles during a qualifying medical procedure.
  Virtual Reality (VR): A child life specialist will fit the patient with the goggles, select a game, and initiate play once the medical procedure begins.
- Standard Care (Control Group): In this arm, patients will receive standard of care with child life specialists during a qualifying medical procedure.
- Reference Group: No virtual reality and no child life specialists; no standardized or formal form of support.
Period: Overall Study
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Started | 19 | 25 | 20
Completed | 17 | 25 | 20
Not Completed | 2 | 0 | 0
Not completed — Procedure cancelled | 1 | 0 | 0
Not completed — VR Malfunction | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Virtual Reality Group (Study Group): In this arm, patients will receive standard of care plus may use virtual reality simulation goggles during a qualifying medical procedure.
  Virtual Reality: A child life specialist will fit the patient with the goggles, select a game, and initiate play once the medical procedure begins.
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group | Total
Number analyzed (Participants) | 17 | 25 | 20 | 62
Age, Customized [Count of Participants; unit: Participants]
  Child (7-9 years) | 3 | 2 | 4 | 9
  Early Adolescent (10-13 years) | 7 | 9 | 3 | 19
  Middle Adolescent (14-17 years) | 6 | 7 | 9 | 22
  Late Adolescent/Adult (18+ years) | 1 | 7 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 12 | 36
  Male | 6 | 12 | 8 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 15 | 23 | 20 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 16 | 11 | 33
  White | 9 | 7 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 25 | 20 | 62
Type of Procedure [Count of Participants; unit: Participants]
  Venipuncture (IV/blood draw) | 17 | 20 | 20 | 57
  Burn debridement | 1 | 1 | 0 | 2
  Laceration repair | 1 | 1 | 0 | 2
  Abscess drainage | 0 | 1 | 0 | 1
  Cast Placement | 0 | 2 | 0 | 2
Child Baseline Pain Level [Mean (Standard Deviation); unit: score on a scale] — Pain described on visual analog scale or Wong-Faces Scale (with a score range of 0-10) with 0 being no pain and 10 being worst pain.
  score on a scale | 4.50 (2.74) | 4.56 (3.73) | 4.75 (3.46) | 4.56 (3.35)
Child Baseline Anxiety Level [Mean (Standard Deviation); unit: score on a scale] — Anxiety described on visual analog scale (0-10), 0 being no anxiety and 10 being worst anxiety.
  score on a scale | 3.94 (2.56) | 3.32 (3.48) | 2.00 (2.79) | 3.03 (3.08)
Adult Baseline Perceived Pain Level [Mean (Standard Deviation); unit: score on a scale] — Pain ratings were based on a 0-10 Likert rating scale with 0 representing the least pain and 10 representing the most. This measure was assessed in caregivers.
  score on a scale | 4.69 (2.68) | 4.95 (3.39) | 5.44 (2.88) | 5.03 (2.99)
Adult Baseline Perceived Anxiety Level [Mean (Standard Deviation); unit: score on a scale] — Anxiety ratings were based on a 0-10 Likert rating scale with 0 representing the least anxiety, and 10 representing the most. This measure was assessed in caregivers.
  score on a scale | 5.25 (2.37) | 4.65 (3.23) | 2.47 (3.71) | 4.21 (3.35)
Adult Baseline Own Anxiety Level [Mean (Standard Deviation); unit: score on a scale] — Anxiety ratings were based on a 0-10 Likert rating scale with 0 representing the least anxiety and 10 representing the most. This measure was assessed in caregivers.
  score on a scale | 4.13 (3.59) | 2.95 (3.12) | 0.47 (1.12) | 2.51 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Pain During the Procedure
Description: Pain described on visual analog scale (0-10), or Wong-Faces Scale (0-10) with 0 being no pain and 10 being worst pain. Change in pain scores (calculated during procedure - pre-procedure) ranges from -10 to 10. A negative number signifies reduced pain during the procedure.
Time Frame: Baseline and Immediately post-procedure, up to 15 minutes
Measure: Mean (Standard Deviation); unit: Visual Analog scale range 0-10
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Visual Analog scale range 0-10 | -0.65 (4.36) | -1.04 (3.86) | 0.95 (2.35)

2. Primary Outcome: Change in Patient-Reported Anxiety During Procedure
Description: Patient anxiety after procedures was described on a visual analog scale (0-10). This is a scale of range 0-10 with 0 being no anxiety and 10 being maximum anxiety. Change in anxiety scores (calculated during procedure - pre-procedure) ranges from -10 to 10. A negative number signifies reduced anxiety during the procedure.
Time Frame: Baseline and Immediately post-procedure, up to 15 minutes
Measure: Mean (Standard Deviation); unit: Visual Analog scale range 0-10
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Visual Analog scale range 0-10 | -0.24 (3.38) | -0.24 (2.76) | 1.45 (3.32)

3. Primary Outcome: Change in Adult Perceived Pain During the Procedure
Description: Perceived pain ratings were obtained for caregivers after the procedure based on a 0-10 Likert rating scale with 0 representing the least pain and 10 representing the most. Change in pain scores (calculated during procedure - pre-procedure) ranges from -10 to 10. A negative number signifies reduced pain during the procedure. This measure was assessed in caregivers.
Time Frame: Baseline and Immediately post-procedure, up to 15 minutes
Measure: Mean (Standard Deviation); unit: Likert rating scale range 0-10
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Likert rating scale range 0-10 | -1.65 (3.35) | -1.70 (3.74) | 0 (2.52)

4. Primary Outcome: Change in Adult Perceived Anxiety During the Procedure
Description: The Subjective Units of Distress scale will be used to measure anxiety of subjects after procedures. This is a scale of 0-10 with 0 being no anxiety and 10 being maximum anxiety. Change in anxiety scores (calculated during procedure - pre-procedure) ranges from -10 to 10. A negative number signifies reduced anxiety during the procedure. This measure was assessed in caregivers.
Time Frame: Baseline and Immediately post-procedure, up to 15 minutes
Measure: Mean (Standard Deviation); unit: Likert scale range 0-10
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Likert scale range 0-10 | -1.12 (4.06) | -1.10 (2.57) | 1.29 (2.47)

5. Primary Outcome: Change in Adult's Own Anxiety During the Procedure
Description: Anxiety ratings were obtained for caregivers after the procedure based on a 0-10 Likert rating scale with 0 representing the least anxiety and 10 representing the most. Change in anxiety scores (calculated during procedure - pre-procedure) ranges from -10 to 10. A negative number signifies reduced anxiety during the procedure. This measure was assessed in caregivers.
Time Frame: Baseline and Immediately post-procedure, up to 15 minutes
Measure: Mean (Standard Deviation); unit: Likert scale range 0-10
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Likert scale range 0-10 | 0.76 (3.85) | -0.95 (2.21) | 0.35 (1.32)

6. Primary Outcome: Child and Adult Medical Procedure Interaction Scale (CAMPIS) Score
Description: Coping was measured using a modified CAMPIS-SF in both patients and caregivers.
  CAMPIS-SF (Child-Adult Medical Procedure Interaction Scale-Short Form) is a behavior rating scale that documents distressing or coping behaviors exhibited in both children and the accompanying adult (parent/guardian). It has been validated to measure coping in children and adults during medical procedures. The CAMPIS-SF study used a 5-point Likert scale to document frequency of each code In order to account for frequency variance due to differences in procedure duration, we used a proportion-based metric validated for CAMPIS-R, and applied this to CAMPIS-SF codes. Proportions were calculated by summing the total number of an event type (e.g. child distress) and dividing by the total number of coded events (child distress plus child coping). This provided a proportion for each event type so that the proportion of child distress plus child coping events add up to 1.0 (range 0-1.0).
Time Frame: Immediately post-procedure, up to 15minutes
Population: 13, 20 and 17 caregivers for the respective arms were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Proportion of total CAMPIS score
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Proportion of total CAMPIS score
  Child Coping Proportion | 0.87 (.18) | .86 (.18) | .70 (.39)
  Child Distress Proportion | 0.13 (.18) | .14 (.18) | .20 (.31)
  Caregiver Coping Proportion: number analyzed (Participants) | 13 | 20 | 17
  Caregiver Coping Proportion | 0.58 (0.39) | .48 (.46) | .57 (.43)
  Caregiver Distress Proportion: number analyzed (Participants) | 13 | 20 | 17
  Caregiver Distress Proportion | .25 (0.30) | .12 (.24) | .20 (.31)

7. Secondary Outcome: Duration of Procedure
Description: Duration of procedure in minutes will be assessed for each procedure.
Time Frame: Immediately post-procedure, up to 20 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
minutes | 13.35 (10.29) | 9.24 (6.58) | 5.1 (4.97)

8. Secondary Outcome: Ease of Procedure as Assessed by a Likert Scale
Description: Ease of procedure will be assessed using a Likert scale completed by proceduralist. The Likert scale ranges from 0-10 with 0 being easy and 10 difficult.
Time Frame: Immediately post-procedure, up to 15 minutes
Measure: Mean (Standard Deviation); unit: Likert scale range 0-10
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Likert scale range 0-10 | 1.4 (2.6) | 0.6 (1.3) | 0.7 (1.3)

9. Secondary Outcome: Personnel Use for Immobilization
Description: This will be assessed using number of patients requiring immobilization during procedures.
Time Frame: Immediately post-procedure, up to 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Participants | 4 | 2 | 0

10. Secondary Outcome: Number of IV or Phlebotomy Attempts
Description: Number of IV or phlebotomy attempts until success will be counted (1 or 2+) in patients undergoing venipuncture procedures.
Time Frame: Immediately post-procedure, up to 15 minutes
Population: This is a sub-analysis of the population undergoing venipuncture procedures only. 5 in the CL group and 2 in the VR group were excluded due to non-venipuncture procedures. 2 patients in the VR group were excluded due to a medical emergency and procedure cancellation.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 15 | 20 | 20
Participants
  1 Attempt | 13 | 16 | 17
  2+ Attempts | 2 | 4 | 3

11. Secondary Outcome: Pre-Procedure Nausea Symptoms
Description: The number of patients reporting nausea symptoms prior to the procedure
Time Frame: Immediately pre-procedure (15minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
Number analyzed (Participants) | 17 | 25 | 20
Participants | 2 | 8 | 4

12. Secondary Outcome: Pre-Procedure Cybersickness Symptoms
Description: Number of patients in the VR group reporting positive cybersickness symptoms prior to the procedure
Time Frame: Immediately pre-procedure (15minutes)
Population: Included patients randomized to VR during the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Group (Study Group)
Number analyzed (Participants) | 17
Participants | 2

ADVERSE EVENTS:
Time Frame: Immediately post-procedure, up to 15minutes.
Description: Symptoms of Cybersickness from the Simulator Sickness Questionnaire. The questionnaire has 16 symptoms with each symptom being scored as present (positive) or absent (negative). Patients with any cybersickness symptoms were designated as 'positive' for cybersickness.
Arm/Group | Virtual Reality Group (Study Group) | Standard Care (Control Group) | Reference Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 3/19 | 4/25 | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Virtual Reality Group (Study Group) (N=19) | Standard Care (Control Group) (N=25) | Reference Group (N=20)
Post-Procedure Nausea (General disorders) | 1 | 4 | 4 — Patients with Post-Procedure Nausea Symptoms
Cybersickness Post-Procedure (General disorders) | 2 | 0 | 0 — Patients with Positive Cybersickness Symptoms Post-Procedure

LIMITATIONS AND CAVEATS:
Early termination due to the COVID-19 pandemic, small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT03686176/Prot_SAP_000.pdf